CLINICAL TRIAL: NCT01054586
Title: HI FPV Study: Using Observational Cohorts to Monitor Safety of Fosamprenavir in Patients With Mild/Moderate Hepatic Impairment
Brief Title: Fosamprenavir in Pts With Hepatic Impairment
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111949; WEUKSTV2430 (Other: GSK); EPI40537 (Other: GSK)
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Results first posted 2011-06-28 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-04

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: antiretroviral therapy; hepatic impairment; HIV
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV pts w/ HBV or HCV, w/ or w/o mild to moderate HI: Patients with HIV coinfected with HBV or HCV with or without mild to moderate HI who are enrolled in one of the participating HIV patient cohorts. These patients will be exposed to FPV/RTV or LPV/RTV.
  Interventions: Drug: Intervention A Standard dose; Drug: Intervention B Reduced Dose; Drug: Intervention C; Drug: Intervention D; Drug: Intervention E

INTERVENTIONS:
Drug: Intervention A Standard dose — HIV subjects with HBV or HCV co-infection but normal hepatic function, defined by receipt of FPV 700mg BID/RTV 100mg BID and a baseline AST-platelet ratio index (APRI) score of <2.0.
Drug: Intervention B Reduced Dose — HIV subjects with mild hepatic impairment, defined by receipt of the recommended reduced FPV/RTV dose (700mg BID/100mg QD).
Drug: Intervention C — HIV subjects with moderate hepatic impairment, defined by receipt of FPV 450mg BID/RTV 100mg QD.
Drug: Intervention D — HIV subjects receiving the standard dose of FPV/RTV despite evidence of abnormal hepatic function according to APRI score: HIV subjects with HBV or HCV co-infection, receipt of FPV 700mg BID/RTV 100mg BID and a baseline APRI score of ≥2.0.
Drug: Intervention E — HIV subjects coinfected with HBV or HCV who have initiated standard doses of LPV 400mg/RTV 100mg and enrolled in the same cohorts as the FPV/RTV exposed subjects.

SUMMARY:
APV10017 was a pharmacokinetic study that evaluated the pharmacokinetics, safety and tolerability of fosamprenavir/ritonavir (FPV/RTV) at reduced doses over 14 days in HIV-infected subjects with mild to moderate hepatic impairment (HI). Based on these data, two new regimens have recently been approved by the EMEA and FDA in these patient groups; FPV 700mg BID/RTV 100mg QD for those with mild HI (Child-Pugh score 4-6) and FPV 450mg BID/RTV 100mg QD for those with moderate HI (Child Pugh score 7-9). The Committee for Medicinal Products for Human Use (CHMP) has requested longer-term safety data among this hepatically impaired HIV-infected population who have received the recently updated FPV/RTV dosing regimens.

An observational cohort study will be conducted using routinely collected data in three European HIV patient cohorts with a high proportion of hepatitis co-infected individuals. Patients who received FPV/RTV will be followed to address the following objectives.

Primary: To assess the safety and tolerability of FPV/RTV-based ART in subjects with mild to moderate hepatic impairment.

Secondary: A). To compare the safety and tolerability of FPV/RTV-based ART in subjects with mild to moderate hepatic impairment when compared to FPV/RTV-based ART in hepatitis B (HBV) or hepatitis C (HCV) co-infected subjects with normal hepatic function. B). To compare the safety and tolerability of FPV/RTV-based ART to lopinavir/ritonavir LPV/RTV-based ART in subjects with mild to moderate hepatic impairment.

DETAILED DESCRIPTION:
Patients were not recruited for nor enrolled in this study. This study is a retrospective observational study. Data from medical records or insurance claims databases are anonymised and used to develop a patient cohort. All diagnoses and treatment are recorded in the course of routine medical practice.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected patients with or without hepatic impairment coinfected with HBV or HCV who started FPV/RTV-based therapy on or after January 1, 2008. The FPV/RTV exposed patients will be stratified into four groups for analysis (see interventions A-D for label/description above), according to their degree of baseline hepatic impairment, which will be defined according to FPV/RTV dose received (and APRI score for interventions A and D). The LPV/RTV intervention group must have started this therapy at approved standard doses on or after January 1, 2008.

Exclusion Criteria:

* Receipt of FPV/RTV or LPV/RTV within the year preceding the baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population is from three HIV patient cohorts; ICONA, HEPAVIH and MASTER cohort in Europe. Data from these cohorts are comprised of the clinical records (or a defined subset thereof) of HIV infected patients. The ICONA Foundation study collects data on HIV infected individuals from 67 infectious disease centres across Italy and has been established since 1997. The ICONA cohort only includes patients who are treatment naïve at initial presentation. HEPAVIH is a cohort of HIV-hepatitis co-infected patients, identified from three other ongoing French HIV cohorts: RIBAVIC, SEROCO and AQUITAINE and an additional 12 clinical departments. The MASTER cohort collects data on HIV infected individuals from centres across Italy and includes treatment-experienced and naive patients.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2009-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As this was an observational, retrospective study, no participants were recruited for participation in this study. For more information about this study, see the protocol in ClinicalTrials.gov and/or search for this study (111949) on http://www.gsk-clinicalstudyregister.com/.
Groups:
- FPV 700 mg BID/RTV 100 mg BID: Fosamprenavir 700 milligrams (mg) twice a day (BID)/Ritonavir 100 mg BID
- FPV 700 mg BID/RTV 100 mg QD: FPV 700 mg BID/RTV 100 mg once a day (QD)
- FPV, Other: All other dosages of FPV (excluding FPV 700 mg BID/RTV 100 mg BID and FPV 700 mg BID/RTV 100 mg QD)
- LPV, Standard Dose: Lopinavir (LPV), Standard Dose
Period: Overall Study
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | FPV, Other | LPV, Standard Dose
Started | 43 | 15 | 8 | 101
Completed | 43 | 15 | 8 | 101
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- FPV, Other: All other dosages of Fosamprenavir
- Total: Total of all reporting groups
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | FPV, Other | LPV, Standard Dose | Total
Number analyzed (Participants) | 43 | 15 | 8 | 101 | 167
Age Continuous [Median (Full Range); unit: years] | 45 [36 to 62] | 45 [29 to 51] | 44 [36 to 53] | 44 [25 to 74] | 44 [25 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 0 | 38 | 52
  Male | 32 | 12 | 8 | 63 | 115
Cohort Distribution [Number; unit: participants] — Source population from three human immunodeficiency virus (HIV)-infected patient cohorts: ICONA (Italian Cohort of Antiretroviral Naïve Patients), treatment naïve participants at initial presentation in Italy; HEPAVIH, HIV-hepatitis coinfected in France; MASTER (Management Standardizzato di Terapia Antiretrovirale), HIV-infected participants who are either treatment experienced or naïve patients in Italy
  participants
    Cohort - MASTER | 36 | 13 | 4 | 72 | 125
    Cohort - HEPAVIH | 3 | 2 | 2 | 6 | 13
    Cohort - ICONA | 4 | 0 | 2 | 23 | 29
Number of participants positive for Hepatitis B and/or C at baseline [Number; unit: participants] — Participant characteristics at baseline according to treatment group. Participants were tested for Hepatitis C antibody (HCV-Ab) and Hepatitis B surface antigen (HBs-Ag).
  participants
    HCV-Ab positive test | 37 | 14 | 7 | 82 | 140
    HBs-Ag positive test | 9 | 2 | 2 | 21 | 34
Number of participants who were ART naïve at baseline [Number; unit: participants] — Participant characteristics at baseline according to treatment group. The number of participants who had not received antiretroviral therapy (ART) was recorded.
  participants | 12 | 5 | 2 | 50 | 69
Number of participants with acquired immunodeficiency syndrome (AIDS) at baseline [Number; unit: participants] — Participant characteristics at baseline according to treatment group. The number of participants with AIDS was recorded.
  participants | 9 | 0 | 3 | 24 | 36
Number of participants with the indicated alanine aminotransferase (ALT) levels at baseline [Number; unit: participants] — Participant characteristics at baseline according to treatment group. The number of participants with the indicated ALT levels was recorded. IU/L = International Units per Liter.
  participants
    Baseline ALT <= 200 IU/L | 40 | 11 | 6 | 83 | 140
    Baseline ALT > 200 IU/L | 1 | 2 | 1 | 3 | 7
    Baseline ALT Unknown | 2 | 2 | 1 | 15 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Events of ALT Elevation After Baseline, Controlling for APRI Score and Other Variables
Description: An elevation in ALT is defined as a single value >200 IU/I.
Time Frame: The incidence of these events was assessed over time during Year 1, censoring participants' follow-up at date of last ALT
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Number; unit: events
Groups:
- ART naïve: Patients that have never been exposed (termed naive) to Antiretroviral (ART) therapy
- Not ART naïve: Patients who have previously been exposed to ART therapy
Arm/Group | ART naïve | Not ART naïve
Number analyzed (Participants) | 69 | 98
events | 9 | 4
Statistical Analysis 1: Comparison: ART naïve vs Not ART naïve; Test type: Superiority or Other; p = 0.02, Regression, Cox — Only variables showing an imbalance between the treatment groups (when possible and besides APRI score) were included. The following were also included, but p > 0.05: APRI score, use of non-ARV drug, baseline CD4, platelets, and bilirubin; Hazard Ratio (HR) = 6.10, 95% CI [1.26 to 29.46] — Confidence Interval and Hazard Ratio for "ART naïve." "Not ART naïve" is the reference group

2. Primary Outcome: Number of Events of an Elevation in ALT After Baseline by Treatment Group, Controlling for APRI-score, and Other Variables
Description: An elevation in ALT is defined as a single value >200 IU/I.
Time Frame: Incidence of these events was assessed over time during Year 1, censoring patients' follow-up at date of last ALT
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Number; unit: events
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | LPV, Standard Dose
Number analyzed (Participants) | 43 | 15 | 101
events | 6 | 1 | 6
Statistical Analysis 1: Comparison: FPV 700 mg BID/RTV 100 mg BID vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.05, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 4.12, 95% CI [1.03 to 16.50] — Confidence Interval and Hazard Ratio for "FPV 700 mg BID/RTV 100 mg BID." "LPV" is the reference group
Statistical Analysis 2: Comparison: FPV 700 mg BID/RTV 100 mg QD vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.68, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.62, 95% CI [0.16 to 16.27] — Confidence Interval and Hazard Ratio for "FPV 700 mg BID/RTV 100 mg QD." "LPV" is the reference group

3. Primary Outcome: Number of Events of an Elevation in ALT After Baseline by Treatment Group, Controlling for FIB-score, and Other Variables
Description: An elevation in ALT is defined as a single value >200 IU/I.
Time Frame: Incidence was assessed over time during Year 1
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Number; unit: events
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | LPV, Standard Dose
Number analyzed (Participants) | 43 | 15 | 101
events | 6 | 1 | 6
Statistical Analysis 1: Comparison: FPV 700 mg BID/RTV 100 mg BID vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.17, Regression, Cox — Only variables showing an imbalance between the treatment groups (when possible) were included. The following were also included, but p > 0.05: APRI score, use of non-ARV drug, baseline CD4, platelets, and bilirubin; Hazard Ratio (HR) = 2.83, 95% CI [0.65 to 12.36] — Confidence Interval and Hazard Ratio for "FPV 700 mg BID/RTV 100 mg BID." "LPV" is the reference group
Statistical Analysis 2: Comparison: FPV 700 mg BID/RTV 100 mg QD vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.85, Regression, Cox — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 1.26, 95% CI [0.12 to 13.33] — Confidence Interval and Hazard Ratio for "FPV 700 mg BID/RTV 100 mg QD." "LPV" is the reference group

4. Primary Outcome: Number of Events of an Elevation in ALT After Baseline by Treatment Group, Controlling for Current Values of CD4 and Platelet Counts
Description: An elevation in ALT is defined as a single value >200 IU/I.
Time Frame: Incidence was assessed over time during Year 1
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Number; unit: events
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | LPV, Standard Dose
Number analyzed (Participants) | 43 | 15 | 101
events | 6 | 1 | 6
Statistical Analysis 1: Comparison: FPV 700 mg BID/RTV 100 mg BID vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.06, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 3.2, 95% CI [0.94 to 10.82] — Confidence Interval and Hazard Ratio for "FPV 700 mg BID/RTV 100 mg BID." "LPV" is the reference group
Statistical Analysis 2: Comparison: FPV 700 mg BID/RTV 100 mg QD vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.96, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.06, 95% CI [0.11 to 9.83] — Confidence Interval and Hazard Ratio for "FPV 700 mg BID/RTV 100 mg QD." "LPV" is the reference group

5. Secondary Outcome: Number of Events of First Discontinuation of FPV/RTV or LPV/RTV Alone by Treatment Group, Controlling for APRI-score, and Other Variables
Description: A first discontinuation is defined as the first occurrence of stopping FPV/RTV or LPV/RTV.
Time Frame: Incidence was assessed over time during Year 1
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Number; unit: events
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | FPV, Other | LPV, Standard Dose
Number analyzed (Participants) | 43 | 15 | 8 | 101
events | 9 | 1 | 4 | 19
Statistical Analysis 1: Comparison: FPV 700 mg BID/RTV 100 mg BID vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.57, Regression, Cox — Variables showing imbalance between treatments (when possible and besides APRI score) were included. Gender, mode of HIV transmission, ART naive, APRI score, use of non-ARV drug, baseline CD4, platelets, and bilirubin were also included, but p>0.05; Hazard Ratio (HR) = 1.31, 95% CI [0.52 to 3.31] — Confidence Interval and Hazard Ratio for "FPV 700 mg BID/RTV 100 mg BID." "LPV" is the reference group
Statistical Analysis 2: Comparison: FPV 700 mg BID/RTV 100 mg QD vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.22, Regression, Cox — [p-value comment as in outcome 5, analysis 1]; Hazard Ratio (HR) = 0.28, 95% CI [0.04 to 2.14] — Confidence Interval and Hazard Ratio for "FPV 700 mg BID/RTV 100 mg QD." "LPV" is the reference group
Statistical Analysis 3: Comparison: FPV, Other vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.47, Regression, Cox — [p-value comment as in outcome 5, analysis 1]; Hazard Ratio (HR) = 1.86, 95% CI [0.35 to 9.91] — Confidence Interval and Hazard Ratio for "FPV, Other." "LPV" is the reference group

6. Secondary Outcome: Number of Events of First Discontinuation of FPV/RTV or LPV/RTV Alone by Treatment Group, Controlling for FIB-score, and Other Variables
Description: A first discontinuation is defined as the first occurrence of stopping FPV/RTV or LPV/RTV.
Time Frame: Incidence was assessed over time during Year 1
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Number; unit: events
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | FPV, Other | LPV, Standard Dose
Number analyzed (Participants) | 43 | 15 | 8 | 101
events | 9 | 1 | 4 | 19
Statistical Analysis 1: Comparison: FPV 700 mg BID/RTV 100 mg BID vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.48, Regression, Cox — Only variables showing imbalance between treatments (when possible) were included. The following were also included, but p > 0.05: gender, mode of HIV transmission, ART naive, APRI score, use of non-ARV drug, baseline CD4, platelets, and bilirubin; Hazard Ratio (HR) = 1.40, 95% CI [0.55 to 3.55] — Confidence Interval and Hazard Ratio for "FPV 700 mg BID/RTV 100 mg BID." "LPV" is the reference group
Statistical Analysis 2: Comparison: FPV 700 mg BID/RTV 100 mg QD vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.23, Regression, Cox — [p-value comment as in outcome 6, analysis 1]; Hazard Ratio (HR) = 0.26, 95% CI [0.03 to 2.18] — Confidence Interval and Hazard Ratio for "FPV 700 mg BID/RTV 100 mg QD." "LPV" is the reference group
Statistical Analysis 3: Comparison: FPV, Other vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.56, Regression, Cox — [p-value comment as in outcome 6, analysis 1]; Hazard Ratio (HR) = 1.67, 95% CI [0.29 to 9.47] — Confidence Interval and Hazard Ratio for "FPV, Other." "LPV" is the reference group

7. Other Pre Specified Outcome: Median Length of Participant Follow-up and Length of Time on Antiretroviral Therapy (ART) at Baseline
Description: Participant characteristics at baseline are presented according to treatment group. ART is used for the treatment of HIV.
Time Frame: Baseline
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Median (Full Range); unit: years
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | FPV, Other | LPV, Standard Dose
Number analyzed (Participants) | 43 | 15 | 8 | 101
years
  Length of follow-up | 0.36 [0.07 to 1.07] | 0.36 [0.04 to 1.02] | 0.95 [0.6 to 1.50] | 0.34 [0.12 to 1.46]
  Tiime on ART | 1.7 [0 to 12] | 1.0 [0 to 11] | 3.21 [0 to 10] | 0.08 [0 to 12.8]

8. Secondary Outcome: Number of Events of First Discontinuation of FPV/RTV- or LPV/RTV Alone by Treatment Group, Controlling for Current Values of CD4 and Platelet Counts
Description: A first discontinuation is defined as the first occurrence of stopping FPV/RTV or LPV/RTV
Time Frame: Incidence was assessed over time during Year 1
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Number; unit: events
Groups:
- FPV 700 mg BID/RTV 100 mg QD: Fosamprenavir 700 mg BID/Ritonavir 100 mg once a day (QD)
- LPV, Standard Dose: Lopinavir, Standard Dose
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | FPV, Other | LPV, Standard Dose
Number analyzed (Participants) | 43 | 15 | 8 | 101
events | 9 | 1 | 4 | 19
Statistical Analysis 1: Comparison: FPV 700 mg BID/RTV 100 mg BID vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.72, Regression, Cox — Only variables showing an imbalance between treatment groups were included: gender, mode of HIV transmission, ART naive, use of non-ARV drug, baseline bilirubin; Hazard Ratio (HR) = 1.16, 95% CI [0.51 to 2.66] — Confidence Interval and Hazard Ratio for " FPV 700 mg BID/RTV 100 mg BID". "LPV" is the reference group
Statistical Analysis 2: Comparison: FPV 700 mg BID/RTV 100 mg QD vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.21, Regression, Cox — [p-value comment as in outcome 8, analysis 1]; Hazard Ratio (HR) = 0.27, 95% CI [0.03 to 2.08] — Confidence Interval and Hazard Ratio for " FPV 700 mg BID/RTV 100 mg QD". "LPV" is the reference group
Statistical Analysis 3: Comparison: FPV, Other vs LPV, Standard Dose; Only variables showing an imbalance between treatment groups were included: gender, mode of HIV transmission, ART naive, use of non-ARV drug, baseline bilirubin; Test type: Superiority or Other; p = 0.15, Regression, Cox; Hazard Ratio (HR) = 2.26, 95% CI [0.74 to 6.97] — Confidence Interval and Hazard Ratio for " FPV, other". "LPV" is the reference group

9. Other Pre Specified Outcome: Cluster of Differentiation (CD4) Count at Baseline
Description: Participant characteristics at baseline according to treatment group. CD4 count is a measurement of how many functional CD4 T-cells are circulating in the blood. The lower the absolute CD4 count, the weaker the immune system.
Time Frame: Baseline
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Median (Full Range); unit: cells/microliter (μl)
Groups:
- FPV 700 mg BID/RTV 100 mg QD: Fosamprenavir 700 mg BID/Ritonavir 100 mg QD
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | FPV, Other | LPV, Standard Dose
Number analyzed (Participants) | 43 | 15 | 8 | 101
cells/microliter (μl) | 355 [66 to 1585] | 331 [113 to 912] | 370 [197 to 427] | 252 [7 to 1113]

10. Other Pre Specified Outcome: Median Aspartate Aminotransferase (AST)-Platelet Ratio Index (APRI) Score at Baseline
Description: The APRI score (AST to platelet ratio index) is an index comprised of biochemical values and is used to determine the degree of hepatic fibrosis. It is calculated as follows: APRI score = ([AST level/Upper Limit Normal]/Platelet counts) x 100. AST = Aspartate aminotransferase. In general, APRI scores range from 0 to >2.0, where scores <0.5 indicate no significant fibrosis, scores >1.5 indicate significant fibrosis, and scores >2.0 have been shown to be best correlated with the presence of cirrhosis.
Time Frame: Baseline
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Median (Full Range); unit: APRI Score
Groups:
- FPV 700 mg BID/RTV 100 mg BID: Fosamprenavir 700 mg BID/Ritonavir 100 mg BID
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | FPV, Other | LPV, Standard Dose
Number analyzed (Participants) | 43 | 15 | 8 | 101
APRI Score | 0.4 [0.06 to 1.73] | 0.53 [0.12 to 3.33] | 0.69 [0.14 to 8.06] | 0.35 [0.06 to 5.04]

11. Other Pre Specified Outcome: Median FIB (a Model of End-stage Liver Disease) Score at Baseline
Description: The FIB-4 score is an index that combines biochemical values (platelets, ALT, AST) and age to determine the degree of hepatic fibrosis. FIB-4 = (Age x AST)/(Platelet counts x ALT1/2). The FIB-4 score ranges between values of 0 to 13. A score of <1.45 indicates no/moderate fibrosis (F0-F1-F2-F3 in the ISHAK classification of fibrosis), whereas a score >3.25 is indicative of extensive fibrosis or cirrhosis (F4-F5-F6). The ISHAK classification of fibrosis is a commonly used scoring system that stages fibrosis from 0-6 (1-2, portal fibrotic expansion; 3-4, bridging fibrosis; 5-6, cirrhosis).
Time Frame: Baseline
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Median (Full Range); unit: FIB Score
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | FPV, Other | LPV, Standard Dose
Number analyzed (Participants) | 43 | 15 | 8 | 101
FIB Score | 0.49 [0.17 to 3.00] | 0.64 [0.18 to 5.87] | 1.96 [0.25 to 13.47] | 0.74 [0.19 to 4.38]

12. Other Pre Specified Outcome: Median Model of End-stage Liver Disease (MELD) Score at Baseline
Description: MELD is a scoring system for assessing the severity of chronic liver disease and is used to predict participant survival. It is calculated using biochemical values as follows: MELD = (0.957 x Log[Creatinine]) + (0.378 x Log[Bilirubin]) + (1.120 x Log[INR]) + 0.6431. INR = International Normalized Ratio for prothrombin time. MELD scores range between 0 and 40, with 40 being the most severe, i.e., 100% mortality. In interpreting the MELD score in hospitalized participants, the 3-month mortality is: score >=40, 100% mortality; 30-39, 83% mortality; 20-29, 76% mortality; 10-19, 27% mortality.
Time Frame: Baseline
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe. MELD scores are not available for the "FPV 700 mg BID/RTV 100 mg QD" group due to missing data.
Measure: Median (Full Range); unit: MELD score
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | FPV, Other | LPV, Standard Dose
Number analyzed (Participants) | 43 | 0 | 8 | 101
MELD score | 5.11 [-4 to 11.85] |  | 6.56 [5.06 to 8.08] | 2.45 [-6 to 22.65]

13. Other Pre Specified Outcome: Median ALT and AST Scores at Baseline
Description: Participants characteristics at baseline according to treatment group.
Time Frame: Baseline
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Median (Full Range); unit: IU/L (International Units per Liter)
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | FPV, Other | LPV, Standard Dose
Number analyzed (Participants) | 43 | 15 | 8 | 101
IU/L (International Units per Liter)
  ALT | 64 [10 to 282] | 53 [28 to 297] | 64 [37 to 568] | 52.5 [7 to 416]
  AST | 52 [16 to 163] | 71 [24 to 291] | 66 [27 to 157] | 45 [16 to 358]

14. Secondary Outcome: Number of Events of First Discontinuation of FPV/RTV or LPV/RTV Alone Due to Adverse Events Only
Description: A first discontinuation is defined as the first occurrence of stopping FPV/RTV or LPV/RTV; where the reason for stopping is attritubed to adverse events only
Time Frame: Incidence was assessed over time during Year 1
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Number; unit: events
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | LPV, Standard Dose
Number analyzed (Participants) | 43 | 101
events | 5 | 7
Statistical Analysis 1: Comparison: FPV 700 mg BID/RTV 100 mg BID vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.10, Regression, Cox; Hazard Ratio (HR) = 3.77, 95% CI [0.79 to 18.05] — Confidence Interval and Hazard Ratio for " FPV 700 mg BID/RTV 100 mg BID". "LPV" is the reference group

15. Secondary Outcome: Number of Events of First Discontinuation of One or More Drugs Included in the FPV/RTV- or LPV/RTV-based Regimen by Treatment Group, Controlling for APRI-score and Other Variables (See Comments)
Description: A first discontinuation is defined as the first occurrence of stopping one or more drugs in the FPV/RTV or LPV/RTV-based regime
Time Frame: Incidence was assessed over time during Year 1
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Number; unit: events
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | FPV, Other | LPV, Standard Dose
Number analyzed (Participants) | 43 | 15 | 8 | 101
events | 16 | 8 | 5 | 24
Statistical Analysis 1: Comparison: FPV 700 mg BID/RTV 100 mg BID vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.02, Regression, Cox — Only variables showing an imbalance between the treatment groups were included, but p > .05: gender, mode of HIV transmission, ART naive, APRI score, baseline use of non-ARV drug, and baseline values of CD4, platelets and bilirubin; Hazard Ratio (HR) = 2.53, 95% CI [1.16 to 5.54] — Confidence Interval and Hazard Ratio for " FPV 700 mg BID/RTV 100 mg BID". "LPV" is the reference group
Statistical Analysis 2: Comparison: FPV 700 mg BID/RTV 100 mg QD vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.05, Regression, Cox — [p-value comment as in outcome 15, analysis 1]; Hazard Ratio (HR) = 4.17, 95% CI [1.54 to 11.27] — Confidence Interval and Hazard Ratio for " FPV 700 mg BID/RTV 100 mg QD". "LPV" is the reference group
Statistical Analysis 3: Comparison: FPV, Other vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.06, Regression, Cox — [p-value comment as in outcome 15, analysis 1]; Hazard Ratio (HR) = 3.67, 95% CI [0.97 to 13.90] — Confidence Interval and Hazard Ratio for " FPV, other". "LPV" is the reference group

16. Secondary Outcome: Number of Events of First Discontinuation of One or More Drugs Included in the FPV/RTV- or LPV/RTV-based Regimen by Treatment Group, Controlling for FIB-score and Other Variables
Description: as for outcome 15
Time Frame: Incidence was assessed over time during Year 1
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Number; unit: events
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | FPV, Other | LPV, Standard Dose
Number analyzed (Participants) | 43 | 15 | 8 | 101
events | 16 | 8 | 5 | 24
Statistical Analysis 1: Comparison: FPV 700 mg BID/RTV 100 mg BID vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.01, Regression, Cox — Only variables showing an imbalance between the treatment groups were included: gender, mode of HIV transmission, ART naive, baseline use of non-ARV drug, and baseline values of CD4, platelets and bilirubin; Hazard Ratio (HR) = 2.68, 95% CI [1.21 to 5.9] — Confidence Interval and Hazard Ratio for " FPV 700 mg BID/RTV 100 mg BID". "LPV" is the reference group
Statistical Analysis 2: Comparison: FPV 700 mg BID/RTV 100 mg QD vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.0004, Regression, Cox — [p-value comment as in outcome 16, analysis 1]; Hazard Ratio (HR) = 4.42, 95% CI [1.61 to 12.08] — Confidence Interval and Hazard Ratio for " FPV 700 mg BID/RTV 100 mg QD". "LPV" is the reference group
Statistical Analysis 3: Comparison: FPV, Other vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.11, Regression, Cox — [p-value comment as in outcome 16, analysis 1]; Hazard Ratio (HR) = 3.07, 95% CI [0.78 to 12.03] — Confidence Interval and Hazard Ratio for " FPV, other". "LPV" is the reference group

17. Secondary Outcome: Number of Events of First Discontinuation of One or More Drugs Included in the FPV/RTV- or LPV/RTV-based Regimen by Treatment Group, Controlling Current Values of CD4 and Platelet Counts
Description: as for outcome 15
Time Frame: Incidence was assessed over time during Year 1
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Number; unit: events
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | FPV, Other | LPV, Standard Dose
Number analyzed (Participants) | 43 | 15 | 8 | 101
events | 16 | 8 | 5 | 24
Statistical Analysis 1: Comparison: FPV 700 mg BID/RTV 100 mg BID vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.03, Regression, Cox — Only variables showing an imbalance between the treatment groups were included: gender, mode of HIV transmission, ART naive, APRI-score, baseline use of non-ARV drug and baseline bilirubin; Hazard Ratio (HR) = 2.09, 95% CI [1.06 to 4.15] — Confidence Interval and Hazard Ratio for " FPV 700 mg BID/RTV 100 mg BID". "LPV" is the reference group
Statistical Analysis 2: Comparison: FPV 700 mg BID/RTV 100 mg QD vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.05, Regression, Cox — [p-value comment as in outcome 17, analysis 1]; Hazard Ratio (HR) = 3.61, 95% CI [1.48 to 8.81] — Confidence Interval and Hazard Ratio for " FPV 700 mg BID/RTV 100 mg QD". "LPV" is the reference group
Statistical Analysis 3: Comparison: FPV, Other vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.10, Regression, Cox — [p-value comment as in outcome 17, analysis 1]; Hazard Ratio (HR) = 2.31, 95% CI [0.85 to 6.32] — Confidence Interval and Hazard Ratio for " FPV, other". "LPV" is the reference group

18. Secondary Outcome: Number of Events of Discontinuation of One or More Drugs in the FPV/RTV- or LPV/RTV Regimen Due to Adverse Events Only
Description: Defined as the occurrence of stopping FPV/RTV or LPV/RTV; where the reason for stopping is attributed to adverse events only
Time Frame: Incidence was assessed over time during Year 1
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Number; unit: events
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | LPV, Standard Dose
Number analyzed (Participants) | 43 | 101
events | 3 | 5
Statistical Analysis 1: Comparison: FPV 700 mg BID/RTV 100 mg BID vs LPV, Standard Dose; Test type: Superiority or Other; p = 0.03, Regression, Cox; Hazard Ratio (HR) = 5.12, 95% CI [1.19 to 22.02] — Confidence Interval and Hazard Ratio for " FPV 700 mg BID/RTV 100 mg BID". "LPV" is the reference group

19. Secondary Outcome: Number of Events of First Discontinuation of FPV/RTV or LPV/RTV Alone Due to the Indicated Adverse Events
Description: Defined as the first occurrence of stopping FPV/RTV or LPV/RTV; where the reason for stopping is attributed to adverse events only. Adverse events can only be attributed to the body system stated (no further specificity is available).
Time Frame: Incidence was assessed over time during Year 1
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Number; unit: events
Groups:
- All Participants: All Participants, across all arms
Arm/Group | All Participants
Number analyzed (Participants) | 167
events
  Hypersensitivity reaction | 1
  GI Tract | 5
  Pancreas | 1
  Nervous system | 2
  Kidneys | 1
  Other side effects (not specified as above) | 3

20. Secondary Outcome: Number of Participants Who Discontinued the Indicated Antiretrovirals for the First Time After Starting FPV/r or LPV/r
Description: Antiretrovirals discontinued for the first time after starting FPV/r or LPV/r
Time Frame: Assessed over time during Year 1
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Number; unit: participants
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | FPV, Other | LPV, Standard Dose
Number analyzed (Participants) | 43 | 15 | 8 | 101
participants
  Ritonavir (full or booster) | 11 | 7 | 2 | 0
  Lopinavir/r | 0 | 0 | 0 | 14
  Fos-amprenavir/r | 3 | 0 | 2 | 1
  Lamivudine | 0 | 0 | 0 | 1
  Abacavir | 0 | 1 | 0 | 1
  Combivir | 0 | 0 | 0 | 2
  Truvada | 2 | 0 | 1 | 3
  Atripla | 0 | 0 | 0 | 2

21. Secondary Outcome: Number of Participants With the Indicated Major Reasons for Discontinuing One or More Drugs in the FPV/r or LPV/r Regimen
Description: Major reasons for discontinuing one or more drugs in the FPV/r or LPV/r regimen
Time Frame: Assessed over time during Year 1
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Number; unit: participants
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | FPV, Other | LPV, Standard Dose
Number analyzed (Participants) | 16 | 8 | 5 | 24
participants
  Virological failure | 0 | 0 | 1 | 0
  Hypersensitivity reaction | 0 | 0 | 0 | 1
  Toxicity - GI tract | 1 | 0 | 0 | 2
  Toxicity - Pancreas | 1 | 0 | 0 | 0
  Toxicity, mainly from nervous system | 1 | 0 | 0 | 0
  Toxicity, mainly from kidneys | 0 | 0 | 0 | 1
  Side effects -any of the above unspecified | 0 | 0 | 0 | 1
  Co-morbidity | 0 | 0 | 2 | 1
  Simplified treatment available | 0 | 0 | 0 | 2
  Structured Treatment Interruption (STI) | 1 | 0 | 0 | 0
  Participant's wish/decision | 0 | 0 | 1 | 3
  Physician's decision | 0 | 0 | 0 | 2
  Non-compliance | 0 | 1 | 0 | 1
  Other causes | 9 | 6 | 0 | 2
  Unknown cause | 3 | 1 | 1 | 8

22. Secondary Outcome: Number of Participants for Which the Reason for Discontinuation of One or More Drugs in the FPV/RTV or LPV/RTV Regimen Was Due to Adverse Events Only
Description: Number of participants for which the reason for discontinuation of one or more drugs in the FPV/RTV or LPV/RTV regimen was due to adverse events only. Adverse events can only be attributed to the body system stated (no further specificity is available)
Time Frame: The incidence of these events was assessed over time during Year 1
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 167
participants
  Hypersensitivity reaction | 2
  GI Tract | 6
  Pancreas | 1
  Nervous system | 2
  Kidneys | 1
  Other side effects (not specified as above) | 3

23. Secondary Outcome: Incidence Rates Per 100 Person-years of Follow-up (PYFU) of Study Main Outcome Measures
Description: Incidence rates per 100 person-years of follow-up of study primary outcome. The numbers analyzed in the category titles represent the number of patients with each event. Incidence rate is the number of new cases per population in a given time period, where the denominator is the sum of the person-time of the at-risk population.
Time Frame: Incidence of these events was assessed over time during Year 1
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Number; unit: incidence rate
Arm/Group | All Participants
Number analyzed (Participants) | 167
incidence rate
  ALT elevations/flares after baseline, n=13 | 18
  1st stop of FPV/RTV or LPV/RTV alone, n=33 | 55
  1st stop >=1 drug in FPV/RTV or LPV/RTV reg., n=53 | 102
  Severe hepatic events, n=0 | 0
  Death or hospitalization due to AIDS, n=1 | 1

24. Other Pre Specified Outcome: Median Blood Platelet Count at Baseline
Description: Participant characteristics at baseline according to treatment group.
Time Frame: Baseline
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Median (Full Range); unit: 10^9/liter
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | FPV, Other | LPV, Standard Dose
Number analyzed (Participants) | 43 | 15 | 8 | 101
10^9/liter | 180 [45 to 327] | 146 [24 to 246] | 145 [44 to 222] | 167 [39 to 396]

25. Other Pre Specified Outcome: Median Bilirubin Level at Baseline
Description: Participant characteristics at baseline according to treatment group.
Time Frame: Baseline
Population: HIV/hepatitis virus co-infected participants enrolled in a number of cohort studies in Europe
Measure: Median (Full Range); unit: milligrams (mg)/deciliter (dl)
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | FPV, Other | LPV, Standard Dose
Number analyzed (Participants) | 43 | 15 | 8 | 101
milligrams (mg)/deciliter (dl) | 0.74 [0.22 to 9.39] | 0.62 [0.42 to 4.3] | 0.83 [0.48 to 29.2] | 0.50 [0.16 to 10]

ADVERSE EVENTS:
Description: This is a retrospective study of pre-existing data; thus, no assessments for Serious or Non-serious Adverse Events were performed.
Arm/Group | FPV 700 mg BID/RTV 100 mg BID | FPV 700 mg BID/RTV 100 mg QD | FPV, Other | LPV, Standard Dose
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.